CLINICAL TRIAL: NCT00294008
Title: Electronic Schizophrenia Treatment Adherence Registry(e-STAR): An Observational, International Study to Evaluate Treatment Adherence in Schizophrenia With Long Acting Risperidone Microspheres
Brief Title: A Study to Evaluate Treatment Adherence in Schizophrenia With Long Acting Risperidone Microspheres (e-STAR)
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR005071
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia; Tranquilizing Agents; Mental Disorders; Therapeutic Uses; Physiological Effects of Drugs; Psychotropic Drugs; Antipsychotic Agents
Keywords: Schizophrenia; Treatment adherence; Antipsychotic agents; Risperidone; Long-acting injectable; Risperdal tablet; Risperidal Consta
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Treatment Adherence and Compliance | interventions — Risperidone

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: Risperdal Consta flexible dosage for 24 months
  Interventions: Drug: Risperdal Consta

INTERVENTIONS:
Drug: Risperdal Consta — flexible dosage for 24 months

SUMMARY:
This study is a non-interventional web based registry designed to assess demographic, treatment and outcomes data in patients receiving treatment with long-acting injectable risperidone. One year retrospective data and 2 year prospective data will be collected.

DETAILED DESCRIPTION:
This study is a multicentre, retrospective and prospective observational, cohort design, determining aggregate drug usage patterns and commonly used clinical outcomes associated with the use of long-acting injectable risperidone. The objectives of this study are to collect sufficient retrospective outcome data to allow the evaluation of treatment outcomes with long acting medication compared to previous treatments and to document clinical effectiveness and long-term treatment outcomes in actual practice. Additional objectives are to prospectively assess medication usage patterns and to evaluate reasons for initiation and/or discontinuation of new antipsychotic medications. The study design is a non-interventional, single-arm, observational survey on the use of long-acting injectable risperidone and other long-acting (depot) or oral atypical antipsychotics, with the aim to assess patient outcomes by existing risk or disease factors, patient characteristics, or previous medication. Having reached agreement with the patient on starting treatment with long-acting injectable risperidone, physicians have the opportunity to document the patient's clinical data in the Registry. At baseline, data will be collected retrospectively over a minimum period of 12-months per patient. Data will be collected prospectively over a 24-month period per patient at approximately 3-month intervals after starting treatment. This study will document data of patients for whom treatment with the new antipsychotic medication is indicated, and who are being treated according to the local label. The start date for collecting data is the date the new antipsychotic treatment is initiated, whether as inpatient or outpatient. The preceding 12 months and the next 2 years are respectively for each patient the retrospective and prospective periods of interest. All patients starting with a new antipsychotic medication, decided after agreement between the physician and the patient, in accordance with the local label, are eligible for inclusion in this survey. While patients participating in randomized clinical trials are not excluded, their participation will be noted. Data will be entered by the treating physician. All data collected must be the result of the normal medical care of the patient. No intervention on treatment decisions permitted. The patient's baseline data will be collected within the first week following initiation of the new antipsychotic treatment. Prospective data collection has to occur 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months and 24 months after initiation of the new antipsychotic treatment. If a patient stops the newly initiated antipsychotic treatment the reason for discontinuation has to be reported. Patients discontinuing newly initiated antipsychotic treatment will continue to be followed for up to 24 months. In retrospective period the following treatment outcomes will be assessed: patient characteristics, treatment history with antipsychotics and other concomitant medication, hospitalization history, reason for initiating the new antipsychotic treatment, treatment satisfaction, remission, clinical global impression (CGI-severity), global assessment of functioning (GAF) and clinical deterioration. In prospective period clinical effectiveness will be assessing the following: employment status, remission, treatment satisfaction, CGI-severity, GAF, clinical deterioration, hospitalization, treatment adherence and (serious) adverse events. Long-acting injectable risperidone is flexible dose (25mg to 75mg), intramuscular injection given into gluteus for 24 months

ELIGIBILITY:
Inclusion Criteria:

* Patients starting treatment with a new antipsychotic medication
* Permitted by their physician to participate in a clinical trial
* Patients with schizophrenia or schizoaffective disorder
* Patients who are an ambulant or not chronically hospitalized for maximal 6 months at the moment of initiation of study
* Patients and/or his/her relative, guardian or legal representative has signed the informed consent form

Exclusion Criteria:

* First antipsychotic treatment ever
* Participating in any other drug study
* Chronically hospitalized and according to physician no possibility of being discharged within the planned observation period
* On clozapine during the last 3 months
* Serious unstable medical condition, including recent and present clinically relevant laboratory abnormalities
* Previous sensitivity history to risperidone and treatment resistant schizophrenia
* Pregnant or breast-feeding female
* Female with planned pregnancy within two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients starting with a new antipsychotic medication, decided after agreement between the physician and the patient, in accordance with the local label, are eligible for inclusion in this survey. While patients participating in randomized clinical trials are not excluded, their participation will be noted.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2004-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the the number of days spent in hospital during the first year with Risperdal Consta compared with the year before Risperdal Consta. | Outcome measure is assessed prospectively over a 24-month period per patient at approximately 3-month intervals after starting treatment. Assessment points are baseline, 3, 6, 9, 12, 15, 18, 21, 24-month.

SECONDARY OUTCOMES:
employment status, remission, treatment satisfaction, CGI-severity, GAF, clinical deterioration, hospitalization, treatment adherence and (serious) adverse events | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24-month

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.